CLINICAL TRIAL: NCT06234891
Title: The Effect of Physiotherapy on Pain, Functionality and Quality of Life Scores in Patients With Chronic Low Back Pain
Brief Title: The Effect of Physiotherapy on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kayseri City Hospital (Other Government)
Responsible Party: Principal Investigator, Havva Talay Çalış, Prof.Dr., Kayseri City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kayseri City Hospital
Record Dates: First submitted 2024-01-21; First posted 2024-01-31 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Chronic Low-back Pain
Keywords: physiotherapy; low back pain; quality of life; functionality
MeSH Terms: conditions — Low Back Pain | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Patients with VAS, ODI and SF-36 quality of life values before treatment, in addition to demographic data, who have applied to our Physical Medicine and Rehabilitation Policlinic in our hospital with chronic low back pain in the last 3 (three) months, are determined, and at least 30 above the age of 18 who received physiotherapy and who did not receive physiotherapy. By calling the patient on the phone and being called to our hospital; patient consents will be obtained and VAS, ODI and SF-36 quality of life values will be questioned.
Who Masked: Outcomes Assessor
Masking Description: Patients in both groups were evaluated after treatment by a physiatrist blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): NSAID
  Interventions: Drug: Nsaid
- Group 2 (Active Comparator): nsaid and physiotherapy
  Interventions: Drug: Nsaid; Other: Phsiotheraphy

INTERVENTIONS:
Drug: Nsaid — Medical treatment
  Other Names: Medical treatment
Other: Phsiotheraphy — Nsaid and phsiotheraphy (hotpack-ultrasound therapy- tens)
  Other Names: Medical treatment and phsiotheraphy
  Arms: Group 2

SUMMARY:
Demographic data of patients diagnosed with chronic low back pain and planned for medical treatment (n:30) and physical therapy in addition to medical treatment (n:30), as well as before and after treatment; Visual analog scale (VAS), Oswestry Disability Index (ODI) and Short form 36 (SF-36) quality of life scoring, Lumbar range of motion (LHA), straight leg raising test (DBK) and hand-finger ground distance (EPZM) were evaluated. Hot pack, transcutaneous electrical nerve stimulation (TENS) and ultrasound were given as physical therapy agents.

DETAILED DESCRIPTION:
Patients with VAS, ODI and SF-36 quality of life values before treatment, in addition to demographic data, who have applied to our Physical Medicine and Rehabilitation Policlinic in our hospital with chronic low back pain in the last 3 (three) months, are determined, and at least 30 above the age of 18 who received physiotherapy and who did not receive physiotherapy.

patient consents obtained and VAS, ODI and SF-36 quality of life values questioned.

Pre- and post-treatment values compared, and intragroup changes compared in both groups and evaluated whether physiotherapy contributes to pain, functionality and quality of life in treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been prescribed medical treatment or physiotherapy for mechanical back pain
* Those with demographic information as well as VAS, ODI information in their files
* Patients between the ages of 20-79 who applied to our hospital with the complaint of chronic low back pain

Exclusion Criteria:

* Non-mechanical back pain
* Patients with physiotherapy contraindications
* Those with inflammatory diseases
* Severe heart failure
* Stroke, spinal cord injury, plegia due to traumatic brain injury
* A history of malignancy
* Active infection during treatment
* Having metal implants in the waist area
* Established osteoporosis
* Those with pacemakers

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog scale (VAS) | at baseline and immediately after treatment
  It is a scale used to evaluate pain intensity. Patients are asked to mark the severity of their pain on a 10 cm line. Patients are asked to mark the place expressing their pain on a line on the scale, where the starting point is no pain and the end point is the most severe pain experienced in life. When calculating, the distance between the marked point and the starting point is measured in cm. An increase in the score means that the severity of pain increases.
Oswestry Disability Index (ODI) | at baseline and immediately after treatment
  It is a valid and reliable scoring in Turkish to evaluate the degree of loss of function in low back pain. It consists of 10 items that question pain severity, self-care, lifting and carrying loads, walking, sitting, standing, sleeping, degree of pain change, travel and social life. Each item is scored between "0" and "5". The maximum score is "100" and the minimum score is "0". The results are evaluated as 0-20 points if it minimally affects daily life, 20-40 points if it is moderate, 40-60 points if it is serious, 60-80 points if it completely restricts it, and 80-100 points if it is bedridden. The disability percentage can be calculated by converting the total score obtained into a percentage system. As the total score increases, the level of disability also increases.

SECONDARY OUTCOMES:
SF 36 | at baseline and immediately after treatment
  Short Form-36 (SF-36) Quality of Life Survey: It is a frequently used survey in studies to evaluate the quality of life. A Turkish adaptation study was conducted and its validity and reliability were demonstrated. It consists of a total of 36 items. SF-36 Quality of Life Questionnaire questions the quality of life considering the last 4 weeks. It has 8 subgroups: physical functions, social functions, role inhibition due to physical problems, physical pain, mental health, role inhibition due to emotional problems, life energy and general health.
range of motion (ROM) | at baseline and immediately after treatment
  Lumbar flexion, extension and lateral flexion ROM measurements were evaluated as limited, painful, open.
Straight leg raising | at baseline and immediately after treatment
  It was considered positive if the patient felt pain between 30-70 degrees when she lifted her leg straight while lying on her back and the knee was at 180 degrees.
Finger-to-ground distance | at baseline and immediately after treatment
  When the patient lumbar flexed forward, the distance between the floor and the ground was measured in centimeters and evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Havva Talay Çalış, Prof, Study Director — Saglik Bilimleri Universitesi
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No